CLINICAL TRIAL: NCT06695494
Title: Enabling Genomic Testing in Cancer of Unknown Primary
Acronym: EGGCUP
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Hoffmann-La Roche (Industry); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp213; ISRCTN42910771 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2024-08-27; First posted 2024-11-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cancer of Unknown Primary; Neoplasm, Unknown Primary
Keywords: Cancer of unknown primary; Cancer
MeSH Terms: conditions — Neoplasms, Unknown Primary; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for genetic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Blood sample collection for gene panel array testing and simultaneous research purposes
  Interventions: Diagnostic Test: Gene panel array; Other: Blood Sample Collection

INTERVENTIONS:
Diagnostic Test: Gene panel array — Blood sample collection for gene panel testing
Other: Blood Sample Collection — Blood sample collection for research purposes

SUMMARY:
Cancer of Unknown Primary (CUP) is where cancer cells are found in the body but the place the cancer began is not known. It is the 6th leading cause of cancer death in the UK and the prognosis is poor with a median survival of 6-9 months. There is a higher than average incidence of CUP in the North West (NW) of England (population of 7.4 million). Precision medicine has transformed treatment strategies in known tumour types, however in CUP there remains an urgent need to better understand CUP molecular characteristics to establish potential roles for novel therapeutic strategies. Treatment options remain limited due to difficulties in determining the primary site of the tumour and the lack of access to validated biomarkers. Access to good-quality tissue for molecular profiling remains a huge challenge in CUP. The emergence of liquid biopsies (sequence DNA in a blood test) as a source of biomarkers is also gaining rapid ground and this study aims to explore the potential utility of liquid biopsies in CUP.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years or over
2. Written informed consent according to ICH/GCP and national regulations
3. ECOG Performance status 0-2
4. Confirmed diagnosis of CUP as per the ESMO guidelines. Patients must have;

   1. The local pathology reports confirming compatibility with CUP diagnosis and the associated slides used for the diagnosis
   2. Discussion at a local CUP MDT confirming diagnosis
5. Availability of archival tumour histological report
6. Willingness to provide blood samples on up to two occasions during the study

Exclusion Criteria:

1. Patient with an immunohistochemistry profile that provides a definitive clinical indication of a primary cancer with a specific treatment
2. Known HIV, Hepatitis B, C positive, due to the difficulties in handling high-risk specimens
3. Patients who are unable to provide fully informed written consent
4. Presence of any medical, psychological, familial or sociological condition that, in the investigator's opinion, will hamper compliance with the study protocol and follow-up schedule
5. Bleeding diathesis (patients' on anticoagulation are permitted to enter the trial if anticoagulation can be safely managed to enable blood sampling)
6. Conditions in which blood sampling may increase risk of complications for the patients and/or investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with cancer of unknown primary
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the utility of cfDNA molecular profiling in patients diagnosed with CUP | 33 months of recruitment + 12 months follow up period or 1 December 2027 whichever comes first
  1. Percentage of patients with adequate cfDNA yields measured using FoundationOne®️ Liquid CDx testing of blood samples obtained at baseline or progression timepoints
  2. Percentage of patients with actionable genomic alterations measured using FoundationOne®️ Liquid CDx testing of blood samples obtained at baseline or progression timepoints
  3. Percentage of patients eligible for personalised treatment options or enrolment on a UK-based clinical trial because of the cfDNA results, measured using FoundationOne®️ Liquid CDx testing of blood samples obtained at baseline or progression timepoints

SECONDARY OUTCOMES:
Data collection repository of readily available information on trails/treatments for patients diagnosed with CUP | 33 months of recruitment + 12 months follow up period or 1 December 2027 whichever comes first
  Develop a data collection repository and readily available information on trials/treatments for patients diagnosed with CUP to be shared at monthly trial management group meetings to ensure that investigators are aware of suitable trial opportunities
Incorporate molecular genomics into routine practice | 33 months of recruitment + 12 months follow up period or 1 December 2027 whichever comes first
  Routinely incorporate molecular genomics as standard of care in patients diagnosed with CUP following FoundationOne®️ CDx or FoundationOne®️ Liquid CDx at baseline and FoundationOne®️ Liquid CDx at progression
Document and feedback genomic results to treating team and patients | 33 months of recruitment + 12 months follow up period or 1 December 2027 whichever comes first
  Documentation and feedback of genomic results/GTAB outcomes to all patients and treating teams following FoundationOne®️ CDx or FoundationOne®️ Liquid CDx at baseline, and FoundationOne®️ Liquid CDx at progression

OTHER OUTCOMES:
Development of novel biomarkers to help in the diagnosis and treatment of patients diagnosed with CUP | Future research sample collection performed at baseline visit. 33 months of recruitment or 1st December 2026 whichever comes first
  Collect samples to be used to investigate novel biomarkers to help in the diagnosis and treatment in patients diagnosed with CUP

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Cook, Principal Investigator — The University of Manchester
Locations (6):
- United Kingdom (6):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, Merseyside
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Northern Care Alliance NHS Foundation Trust, Manchester
  - University Hospitals of Morecambe Bay NHS Trust, Morecambe
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston